CLINICAL TRIAL: NCT02610491
Title: The Effect of Hesperidin Administration on Glucose / Insulin Metabolism
Brief Title: The Effect of Hesperidin on Glucose / Insulin Metabolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Bouke Salden, MD, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 143036
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — Hesperidin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Cellulose
  Interventions: Dietary Supplement: Placebo
- Hesperidin (Active Comparator): Citrus peel extract
  Interventions: Dietary Supplement: Hesperidin

INTERVENTIONS:
Dietary Supplement: Hesperidin — Citrus peel extract
  Arms: Hesperidin
Dietary Supplement: Placebo — Cellulose
  Arms: Placebo

SUMMARY:
Metabolic Syndrome (MS) is a well-known group of obesity-related metabolic disorders including insulin resistance (IR), dyslipidemia and hypertension (HTN). In addition, overweight has a causal relationship with a chronic low grade systemic inflammatory condition and increased intestinal permeability. Over the last decade, this multiplex disorder has progressively become a major worldwide public health problem, because of its association with increased risk of type 2 diabetes mellitus (DM2), atherosclerotic cardiovascular disease and all-cause mortality. Scientific evidence for measures to improve cardiometabolic and intestinal health by non-pharmaceutical means are of urgent need. Administration of the flavonoid hesperidin to those at risk may have beneficial effects on glucose / insulin metabolism, lipid metabolism, blood pressure, heart rate, pro-inflammatory and oxidative stress biomarkers and gut barrier function.

Objective: To determine the 12-week effect of daily administration of hesperidin on the main cardiometabolic disorders related to MS as assessed by investigation of glucose/insulin metabolism, blood lipid profile, blood pressure, heart rate, body composition and gut barrier function in subjects at risk for MS.

Study design: This is a randomized, double-blind, placebo-controlled study with parallel design.

Study population: Healthy (male/female) volunteers, age 18-65, at risk for metabolic syndrome (presenting with 2 out of 5 of the components from NCEP-ATP-III criteria).

Intervention: Participants will be randomly assigned to one of the intervention groups. One group will receive one daily dose of hesperidin capsules while the other group receives identical looking placebo capsules for a period of 12 weeks. The capsules will have to be ingested with a glass of water every morning just before breakfast.

Main study parameters/endpoints: The primary efficacy parameter of this study is the oral glucose tolerance test (OGTT), a validated surrogate endpoint to study the β-cell function and insulin sensitivity. Secondary endpoints entail the evaluation of effects of daily administration of hesperidin on lipid profile (blood measurements), blood pressure and heart rate, body composition, low-grade inflammation biomarkers (blood measurements) and gut barrier function (blood measurements, fecal samples, urine collection).

ELIGIBILITY:
Inclusion Criteria:

* Subjects at risk for metabolic syndrome: a combination of 2 out of 5 components:

* Waist circumference: men > 102 cm / women > 88 cm
* Triglycerides: ≥ 1.7 mmol/l
* HDL-cholesterol: men ≤ 1.0 mmol/l / women ≤ 1.3 mmol/l
* Systolic blood pressure: ≥ 130 mmHg or diastolic blood pressure: ≥ 85 mmHg
* Fasted serum glucose ≥ 6.1 mmol/L

Exclusion Criteria:

* Type 2 diabetes mellitus (defined as fasting plasma glucose ≥7.0 mmol/l)
* Gastroenterological diseases or abdominal surgery
* Cardiovascular diseases, cancer, liver or kidney malfunction, thyroid disorders, disease with a life expectancy shorter than 5 years
* Self-admitted HIV-positive status
* Abuse of products; alcohol (> 20 alcoholic consumptions per week) and drugs
* Smoking
* Plans to lose weight or following a hypocaloric diet during the study period
* Weight gain or loss > 3 kg in previous 3 months
* Use of medication interfering with endpoints
* Use of antioxidants, minerals and vitamin supplements available in pharmacies, drugstores, food markets or in alternative medicine
* Hormone replacement therapy (women).
* Use of antibiotics in the 90 days prior to the start of study
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator) in the 180 days prior to the study
* Known pregnancy (assessed by a pregnancy test before start of study) or lactation
* Blood donation within 3 months before study period
* Failure to comply prohibited intake of hesperidin containing food products during study period. A list with forbidden products will be provided to participants
* History of any side effects towards the intake of flavonoids or citrus fruits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effect on blood glucose concentrations measured by oral glucose tolerance test | 12 weeks

SECONDARY OUTCOMES:
Effect on blood lipid profile | 12 weeks
Effect on blood pressure | 12 weeks
Effect on body composition measured by BMI | 12 weeks
Effect on low-grade inflammation measured by blood concentration of TNFalfa | 12 weeks
Effect on low-grade inflammation measured by blood concentration of interleukin-6 | 12 weeks
Effect on gut barrier function measured by a sugar test | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MUMC+, Maastricht, Limburg, Netherlands